CLINICAL TRIAL: NCT01183078
Title: Distal Locking Using an Electromagnetic Field Guided Computer Based Real Time System for Orthopaedic Trauma Patients
Acronym: Sure Shot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00012034
Record Dates: First submitted 2010-08-11; First posted 2010-08-17 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2018-07

CONDITIONS: Tibial Fractures; Femoral Fractures
Keywords: efficacy; drill placement; nail placement; radiation; Operative time; Reduction in exposure to radiation; Accuracy for nail placement
MeSH Terms: conditions — Tibial Fractures; Femoral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free-hand technique (Other): Free-hand technique utilized to find screw holes.
  Interventions: Procedure: free-hand
- Wand technique (Other): Wand technique is utilized to find screw holes.
  Interventions: Procedure: Wand technique

INTERVENTIONS:
Procedure: free-hand — Free-hand technique utilizes x-rays to find screw holes.
  Arms: Free-hand technique
Procedure: Wand technique — Wand technique is utilized to find screw holes.
  Arms: Wand technique

SUMMARY:
Hypothesis: Utilization of the "wand" method will enhance improvements in drill placement, locking nail placement during tibia and femur fracture repairs, and offer less radiation exposure and less operative time. The purpose of this research study is to compare the efficacy of distal locking of intramedullary nails using a standard free-hand technique with the guided wand technique. Distal locking is the placement of screws through the intramedullary rod to hold it in place and prevent rotation. Currently, the free-hand technique is most often utilized. With this technique, the surgeon uses intraoperative x-rays in order to find the holes in the intramedullary rod to place the screws. The wand technique uses electromagnetic fields rather than x-rays to find these screw holes. The utilization of the wand technique could result in improvements in drill placement and locking nail placement as well as decrease operative time and radiation exposure.

DETAILED DESCRIPTION:
Methods and Measures Patients 18 years of age and older presenting through the emergency room at Wake Forest University Baptist Medical Center with tibial and femoral fractures suitable for operative repair will be prospectively enrolled. Inclusion criteria will include any patient with a tibia fracture or femur fracture requiring intramedullary nailing. Retrograde intramedullary nails will be excluded as will nails which are not interlocked. The goal for enrollment is 24 tibial and 24 femoral fractures. Data including operative time, C-arm time, and "nail misses" will be obtained in the operating room for 24 tibial and 24 femoral nails. Surgeons who perform the procedure will have had experience using the freehand technique and will be trained with the guided wand prior to the experiment. Locking will be performed with the freehand and the wand technique in alternating order for the two interlocking screws. The order of which technique is utilized first will be randomly assigned. All procedures will be timed, and fluoroscopy time, radiation time, and any "nail misses" will be documented. All tibial nails will be locked with 2 mediolateral screws and all femurs with 2 lateral to medial screws.

Patients will receive follow-up for complications for a 6 month period after surgical procedure. Intervals of follow-up will be at 2 weeks, 6 weeks, 3 months and 6 months. Anterior-posterior and lateral images will be performed as are already customary and usual at these time intervals.

Outcome Measure(s) The goal is to prospectively assess the "wand" technique as a reliable alternative to standard interlocking screw placement which reduced operative time, C-arm exposure and inadvertent "nail misses." Additionally, it is expected that there will exist no complications related to the use of this technique.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older with tibial or femoral fracture suitable for operative repair with intramedullary nailing.

Exclusion Criteria:

* Fractures requiring repair by retrograde intramedullary nails and interlocking nails.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Reduced operative time. | Six months post surgery
  The goal is to prospectively assess the "wand" technique as a reliable alternative to standard interlocking screw placement which reduces operative time.
Reduced C-arm exposure | Six months post surgery
  The goal is to prospectively assess the "wand" technique as a reliable alternative to standard interlocking screw placement, which reduces C-arm exposure.
Reduces inadvertent nail misses. | Six months post surgery
  The goal is to prospectively assess the "wand" technique as a reliable alternative to standard interlocking screw placement, which reduces inadvertent "nail misses."
No complications | Six months post surgery
  The goal is to prospectively assess the "wand" technique as a reliable alternative to standard interlocking screw placement. It is expected that there will exist no complications related to the use of this technique.

CONTACTS AND LOCATIONS:
Overall Officials: Riyaz H. Jinnah, MD, FRCS, Principal Investigator — Wake Forest University Health Sciences; Eben A. Carroll, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences - CompRehab, Winston-Salem, North Carolina, United States